CLINICAL TRIAL: NCT04871100
Title: Addressing Mental Health Comorbidities: Integrated CBT to Improve Functioning in Veterans With Co-Occurring Anxiety and Substance Use
Brief Title: Integrated CBT to Improve Functioning in Veterans With Anxiety and Substance Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3520-W; 1IK2RX003520-01A2 (NIH)
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorder; Posttraumatic Stress Disorder; Hazardous Drinking
Keywords: Veterans; anxiety; Stress Disorders, Post-Traumatic; Alcohol Drinking; psychosocial functioning
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the intervention or a control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UP-A (Experimental): Cognitive behavior therapy using the Unified Protocol for Emotional Disorders with supplemental skills-based alcohol modules.
  Interventions: Behavioral: Unified Protocol- Alcohol
- Enhanced Usual Care (Active Comparator): referrals to VA care for SUD and anxiety
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Unified Protocol- Alcohol — Transdiagnostic cognitive behavior therapy for emotional disorders modified to include CBT for alcohol use.
  Arms: UP-A
Behavioral: Usual care — referrals to VA care for SUD and anxiety
  Arms: Enhanced Usual Care

SUMMARY:
Individual with anxiety and post-traumatic stress disorder often use alcohol in ways that could cause them harm. Treating both mental health concerns and alcohol use at the same time can help reduce difficulties engaging in multiple treatments. The investigators are evaluating how a cognitive behavioral therapy program that helps Veterans with anxiety, posttraumatic stress disorder, and alcohol use at the same time can help improve the participants lives.

DETAILED DESCRIPTION:
Co-occurring hazardous drinking, anxiety disorders, and PTSD are problematic combinations of mental health concerns experienced by deployed Veterans. Veterans who have been deployed are at particular risk for experiencing problems in functioning and reintegration related to mental health disorders and hazardous drinking. Co-occurring anxiety and hazardous drinking heavily impact psychosocial functioning and quality of life. Although cognitive behavior therapy (CBT) can promote psychological recovery through improvements in functioning and quality of life, most CBT protocols do not address co-occurring disorders, leading to inefficient and disjointed treatment. The current research seeks to adapt and test the Unified Protocol (UP) for deployed Veterans with hazardous drinking. The use of combined CBT for both anxiety disorders and hazardous drinking has the potential to more efficiently and effectively improve functioning, reduce symptoms, and promote psychosocial recovery.

ELIGIBILITY:
Inclusion Criteria:

* meeting diagnostic criteria for current anxiety disorder and
* endorsing hazardous alcohol use

Exclusion Criteria:

-need for acute medically-supervised detoxification with exclusionary criteria of

* high-risk suicidality
* psychotic symptoms, or
* cognitive impairment that could interfere with engagement in weekly psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Social Adjustment Scale- Self Report | 2-weeks
  Evaluates individuals' satisfaction with social situation. Greater scores reflect greater social/occupational impairment (range 42-210).
Beck Anxiety Inventory | past 30 days
  Evaluates levels of anxiety in past month. Higher scores reflect greater anxiety (range 0-63).
Addiction Severity Index | 30 days
  Assessment of substance use and related problems. Higher scores in each domain indicate problems related to substance use in that domain (range for each domain 0-1).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Ecker, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ecker AH, Amspoker AB, Johnston W, Walder A, Lindsay JA, Hogan JB. The role of depression and anxiety symptom severity in remotely delivered mental health care. Psychol Serv. 2024 Feb;21(1):42-49. doi: 10.1037/ser0000775. Epub 2023 Jun 22. PMID 37347915
- [Result] Ecker AH, Cucciare MA, Lindsay JA. Overcoming barriers to care for Alcohol Use Disorder: Pathways for change. J Hosp Med. 2025 May;20(5):528-529. doi: 10.1002/jhm.13554. Epub 2024 Nov 14. No abstract available. PMID 39542875
- [Result] Haskins C, Amspoker AB, Walder A, Hogan J, Ecker A, Lindsay J, Shore J. Telehealth Buprenorphine Initiation for Opioid Use Disorder Among American Indian and Alaska Native Veterans, April 2017-March 2023. Telemed J E Health. 2025 Nov;31(11):1333-1341. doi: 10.1089/tmj.2025.0038. Epub 2025 Jul 10. PMID 40637596